CLINICAL TRIAL: NCT06100224
Title: Piloting a Healthy Aging Cohort in Manitoba - PACMan
Brief Title: Piloting a Healthy Aging Cohort in Manitoba
Acronym: PACMan
Status: Recruiting | Type: Observational
Sponsor: University of Manitoba (Other)
Collaborators: Seven Oaks Hospital Chronic Disease Innovation Centre (Network); The Wellness Institute Powered by Seven Oaks General Hospital (Unknown); Medical Fitness Association (Unknown)
Responsible Party: Principal Investigator, Claudio Rigatto, Professor of Medicine, Nephrologist, University of Manitoba
Other Study IDs: HS25790 (H2022:393)
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Healthy Aging
Keywords: Medical fitness facility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to set up and pilot baseline data collection for a prospective cohort designed to explore the relationships between medical fitness facility usage, lifestyle behaviours and health outcomes as individuals age. Additionally, this pilot study will set up the overall objectives for the larger, prospective cohort study using a public engagement participatory approach with public/patient partners involved in determining which healthy aging outcomes to include.

DETAILED DESCRIPTION:
This project will cover the set-up, development, and user-testing of the baseline visit data collection in the first 100 participants. Data will be collected on physical activity, diet, sleep, stress, cognition, frailty, health history (including diabetes, alcohol and smoking), facility and program usage at the Wellness Institute (WI), height, weight, volitional oxygen intake (VO2 max), blood pressure, heart rate, clinical chemistry, urinalysis, body composition, social determinants of health, and wellbeing.

Additionally, a public engagement participatory approach will be used to determine which healthy aging outcomes are important to study, including discussion on research priorities, research question, research design, data collection approaches, outcome measures, analysis of results, relevance of findings, and dissemination of findings. Therefore, this pilot project will include the formation of a project advisory group that will include public/patient partners. The advisory group members will discuss ideas around healthy aging and lifestyle and what outcomes are most important to them; and will provide information on the reasons for joining as well as the use of the medical fitness facility, any barriers they face and program needs. The project advisory group will be an integral part of this pilot project. The information obtained from the advisory group meetings and the pilot project will be used to develop the outcomes for the larger cohort study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 30 years or above.
* Able to communicate in English and provide written informed consent
* Current member of the Wellness Institute
* Access to a device such as an android or iOS smartphone or tablet for use with the dietary tracking application.

Exclusion Criteria:

* Female participant who is pregnant or lactating
* Employees of the Wellness Institute
* Involvement in the planning and/or conduct of the study

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from individuals that attend The Wellness Institute. This study is a pilot with the number of recruited participants set as the initial 20 plus an additional anticipated 80, totaling 100 participants.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Health History | At baseline an Year 1
  Collected using the Chronic Conditions, Health History and Facility Usage Questionnaire and the Family Medical History Questionnaire
Fitness Level | At baseline an Year 1
  Measured by volitional oxygen intake, otherwise known as VO2 max, using the Ebbeling Treadmill Test (a submaximal walking test)
Diet | At baseline an Year 1
  Measured using the Mindful Eating Questionnaire and the 3 Factor Eating Questionnaire
Dietary Intake | At baseline an Year 1
  The RxFood App will be used to measure dietary intake over 3 full days.
Physical Activity | At baseline an Year 1
  Measured using the International Physical Activity Questionnaire - Short form (IPAQ-S)
Physical Activity Assessment | At baseline an Year 1
  An Actigraph activity monitor will be used to measure physical activity for 7 days, wtih participants asked to wear the monitor at all times.
Sleep Quality Assessment | At baseline and Year 1
  Measured using the Pittsburgh Sleep Quality Index Questionnaire (PSQI), an effective instrument used to measure the quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep quality by measuring seven areas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medications, and daytime dysfunction.
Sleep Assessment | At baseline and Year 1
  An ActiGraph activity monitor will be used to measure sleep quality patterns for 7 days, wtih participants asked to wear the monitor at all times, including when they sleep.
Stress | At baseline and Year 1
  The Perceived Stress Questionnaire (PSQ) will be completed to assess stressful life events and circumstances that tend to trigger or exacerbate disease symptoms.
Cognition Assessment | At baseline and Year 1
  The Montreal Cognitive Assessment Score (MoCA) will be used to give insight into how participants mentally process information.
Body Weight | At baseline and at Year 1
  Body weight will be measured.
Body Mass Index (BMI) | At baseline and at Year 1
  Body Mass Index will be measured
Waist circumference | At baseline and at Year 1
  Waist circumference will be measured
Blood Pressure | At baseline and at Year 1
  Blood pressure while awake, while asleep, and total will be measured using an ambulatory blood pressure monitor, worn for 3 consecutive days.
Frailty | At baseline and at Year 1
  The Short Physical Performance Battery (balance test, gait speed, and chair stand) and handgrip strength with be collected to measure frailty.
Facility Usage | At baseline and at Year 1
  Participants will complete a questionnaire on attendance in hours per week, and # of times per week, and specific program/facility usage at the Wellness Institute. The Wellness Institute swipe data will be used to record the number of times swiped per week and per month since joining.
Cholesterol | At baseline and at Year 1
  Total cholesterol, HDL-C, LDL-C, triglycerides, total cholesterol/HDL ratio
HbA1c | At baseline and at Year 1
  Hemoglobin A1C
eGFR | At baseline and at Year 1
  Estimated glomerular filtration rate.
uACR | At baseline and at Year 1
  Urine albumin to creatinine ratio
10-Year Risk of Cardiovascular Disease | At baseline and at Year 1
  Measured using the Framingham Risk Score
Cardiovascular Assessment | At baseline and at Year 1
  Identification of Metabolic Syndrome and the Framingham Risk Score will be measured.
Body Composition | At baseline and at Year 1
  DEXA scan measurements including total mass, fat mass, lean mass, % fat, visceral adipose tissue, total body bone mineral density), and relative skeletal muscle index (RSMI) will be collected.
Social Determinants of Health | At baseline and at Year 1
  Access to general medical and dental care, postal code, household income, education level and marital status will be collected.
Wellbeing - Quality of Life | At baseline and at Year 1
  the EQ-5D-5L will be collected to measure quality of life.
Wellbeing - Loneliness | At baseline and at Year 1
  The UCLA Loneliness Scale will be sued to measure loneliness.
Wellbeing - Life Satisfaction | At baseline and at Year 1
  The Satisfaction With Life Scale will be used to measure life satisfaction
Wellbeing - Self-efficacy | At baseline and at Year 1
  The Multidimensional Health Locus of Control (MHLC) Scale Form A will be used to measure self-efficacy
Wellbeing - Depression | At baseline and at Year 1
  The Center for Epidemiologic Studies Short Depression Scale (CES-D-10) will be used to measure depression

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Rigatto, MD, Principal Investigator — University of Manitoba
Locations (1):
- Seven Oaks Hospital Chronic Disease Innovation Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided